CLINICAL TRIAL: NCT00021112
Title: Surgical Treatment Of Stage IIIB Non-Small Cell Lung Cancer After Induction-Chemoradiotherapy
Brief Title: Combination Chemotherapy Plus Radiation Therapy Followed by Surgery in Treating Patients With Stage IIIB Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-08981; EORTC-08981
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy and radiation therapy before surgery in treating patients who have stage IIIB non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence of radically resected disease in patients with stage IIIB non-small cell lung cancer treated with induction cisplatin, etoposide, and radiotherapy followed by surgical resection.
* Determine the toxicity (morbidity and mortality) of this regimen in these patients.
* Determine the clinical response rate and pathological response rate in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive induction chemotherapy comprising cisplatin IV on day 1 and etoposide IV on days 1-3. Chemotherapy repeats every 3 weeks for 3 courses. Beginning on day 2 of the second course of chemotherapy, patients undergo induction radiotherapy once daily 5 days a week for 5-7 weeks. Chemoradiotherapy continues in the absence of disease progression or unacceptable toxicity.

At 3-6 weeks after completion of the last dose of induction radiotherapy, patients undergo lobectomy or pneumonectomy.

Patients are followed at 30 days and 4 months, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 27-62 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary stage IIIB non-small cell lung cancer (NSCLC)

  * T4, any N, M0 or any T, N3, M0
  * No N3 disease due to scalene or supraclavicular lymph node involvement
* No primary tumors located in the lower lobe combined with contralateral upper higher mediastinal lymph node involvement
* No mixed tumor types with small cell lung cancer
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
* No pre-existing pleural or pericardial effusion
* No CNS involvement by CT scan or MRI

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm ^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.25 times ULN
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No clinical evidence of superior vena cava syndrome

Pulmonary:

* Postoperative FEV1 and KCO greater than 40% predicted
* VO2 max greater than 15 mL/min/kg (if postoperative KCO no greater than 40% predicted)

Other:

* No other primary malignancy except carcinoma in situ of the cervix, adequately treated basal cell skin cancer, or other malignancy treated more than 5 years ago without recurrence (excluding melanoma, breast cancer, or hypernephroma)
* No active uncontrolled infection requiring IV antibiotics
* No pre-existing sensory neurotoxicity grade 2 or greater
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for NSCLC
* No concurrent immunotherapy during induction chemoradiotherapy
* Concurrent colony stimulating factors allowed

Chemotherapy:

* No prior chemotherapy for NSCLC

Endocrine therapy:

* No concurrent anticancer hormonal agents (except corticosteroids for antiemetic prophylaxis) during induction chemoradiotherapy

Radiotherapy:

* No prior radiotherapy for NSCLC

Surgery:

* No prior surgery for NSCLC

Other:

* No other concurrent anticancer drugs during induction chemoradiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2001-04; Primary Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Van Klaveren, MD, PhD, Study Chair — University Medical Center Rotterdam at Erasmus Medical Center
Locations (10):
- Belgium (2):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Universitair Ziekenhuis Antwerpen, Edegem
- Thoraxklinik Rohrbach, Heidelberg, Germany
- Netherlands (5):
  - Gelre Ziekenhuizen - Lokatie Lukas, Apeldoorn
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Rotterdam Cancer Institute, Rotterdam
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Poland (2):
  - Medical University of Gdansk, Gdansk
  - National Institute of Tuberculosis and Lung Diseases, Warsaw